CLINICAL TRIAL: NCT01667523
Title: The Effect of Capsaicin and Cinnamaldehyde on Intestinal Permeability, Gallbladder Motility and Satiety
Brief Title: The Effect of Capsaicin and Cinnamaldehyde on Intestinal Permeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Gastro, Professor Ad. AAM Masclee, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MEC 10-3-058
Record Dates: First submitted 2011-04-12; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: capsaicin; cinnamaldehyde
MeSH Terms: interventions — Capsaicin; cinnamaldehyde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Capsaicin (Experimental)
  Interventions: Dietary Supplement: Capsaicin
- Cinnamaldehyde (Experimental)
  Interventions: Dietary Supplement: Cinnamaldehyde
- Placebo (Placebo Comparator): Physiological saline
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Capsaicin — 1.5 mg capsaicin administered intraduodenally
  Arms: Capsaicin
Dietary Supplement: Cinnamaldehyde — 70 mg per intervention administered intraduodenally
  Arms: Cinnamaldehyde
Dietary Supplement: Placebo — Physiological saline
  Arms: Placebo

SUMMARY:
An altered permeability has been proposed to play an important role in the pathogenesis of several gastrointestinal disorders, such as irritable bowel syndrome and inflammatory bowel disease. Nutrients derived from food are able to influence the permeability of the intestine and can therefore also affect gastrointestinal symptoms. In this study, the investigators will investigate the effects of capsaicine and cinnamaldehyde, which can be found in hot peppers and cinnamon, respectively, on gastrointestinal physiology.

Objective:

To obtain more information about the effects of capsaicin and cinnamaldehyde on the intestine, these substances will be infused directly in the duodenum. Hereafter, the permeability of the intestine, gallbladder motility and the effects on satiety will be assessed.

Hypothesis:

Duodenal capsaicin and cinnamaldehyde infusion induces changes in the intestinal epithelial barrier function by selectively acting on TRPV1 and TRPA1 receptors and releasing serotonin from enterochromaffin cells as determined by the multi sugar permeability test

ELIGIBILITY:
Inclusion Criteria:

1. Based on medical history and previous examination, no gastrointestinal complaints can be defined.
2. Age between 18 and 65 years. This study will include healthy adult subjects. Subjects over 65 years have an increased risk for comorbidities, therefore, subjects over 65 years will not be included. Furthermore, age has an influence on the homeostasis of the intestinal mucosa [21], which can potentially influence outcome parameters of the study.
3. BMI between 20 and 30 kg/m2

Exclusion Criteria:

1. History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
2. Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
3. Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
4. Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
5. Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic), pregnancy, lactation
6. Excessive alcohol consumption (>20 alcoholic consumptions per week)
7. Smoking
8. Blood donation within 3 months before the study period
9. Self-admitted HIV-positive state

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of capsaicin and cinnamaldehyde (CA) infusion on intestinal permeability | Measured at start and end of infusion (30 min), on each of the 3 test days
  Measurements performed in plasma

SECONDARY OUTCOMES:
To assess the effect of capsaicin and CA infusion on the activation of the TRP receptors as defined by the mucosal concentrations of the neuropeptides SP, CGRP and NKA | 1 day
  Measurements will be performed in mucosal biopsy samples
To assess the effect capsaicin and CA on parameters that are known to be associated with satiety, measured by satiety hormones in blood plasma and mucosal tissue (CCK) as well as satiety scoring on a visual analogue scale | 1 day
  Visual analogue scores will be collected from the start of the infusion until 90 minutes thereafter.
To assess the effect of capsaicin and CA on serotonergic function in duodenal biopsy specimens by measuring serotonin and its metabolites by HPLC | 1 day
  Measurements will be performed on biopsy specimens
To assess the effect of capsaicin and CA on gallbladder motility by ultrasound | Measurements will be performed during the testday starting from 08.00 AM to 11.00AM
To assess the effect of capsaicin and CA on the expression of tight junction proteins measured by immunohistochemistry and by quantitative PCR | 1 day
  Measurements will be performed in biopsy specimens of the duodenal mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van Avesaat M, Troost FJ, Westerterp-Plantenga MS, Helyes Z, Le Roux CW, Dekker J, Masclee AA, Keszthelyi D. Capsaicin-induced satiety is associated with gastrointestinal distress but not with the release of satiety hormones. Am J Clin Nutr. 2016 Feb;103(2):305-13. doi: 10.3945/ajcn.115.123414. Epub 2015 Dec 30. PMID 26718419